CLINICAL TRIAL: NCT07330297
Title: The Capabilities of Exhaled Breath Mass Spectrometry in Identifying Metabolic Syndrome and Metabolically Healthy Obesity
Brief Title: Breath Mass Spectrometry in Metabolic Syndrome and Metabolically Healthy Obesity
Status: Recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MHO-MetS-Breath-001
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Syndrome; Obesity & Overweight; Metabolically Healthy Obesity
Keywords: Breath Analysis; Volatile Organic Compounds; Proton-Transfer-Reaction Mass Spectrometry; Artificial Intelligence; Machine Learning; Metabolic syndrome; Obesity; Metabolically healthy obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Overweight; Obesity, Metabolically Benign

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metabolic Syndrome Group: 100 patients diagnosed with Metabolic Syndrome according to International Diabetes Federation (IDF) 2006 criteria.
  Interventions: Diagnostic Test: Breath Sampling and Analysis by PTR-MS
- Metabolically Healthy Obesity Group: 100 patients with waist circumference ≥94 cm (men)/≥80 cm (women), but without other components of Metabolic Syndrome (hypertension, dyslipidemia, impaired fasting glucose).
  Interventions: Diagnostic Test: Breath Sampling and Analysis by PTR-MS
- Control Group: 100 individuals with normal BMI and no signs of Metabolic Syndrome.
  Interventions: Diagnostic Test: Breath Sampling and Analysis by PTR-MS

INTERVENTIONS:
Diagnostic Test: Breath Sampling and Analysis by PTR-MS — A single sample of exhaled breath will be collected from each participant during quiet breathing. The sample will be analyzed in real-time using Proton-Transfer-Reaction Time-of-Flight Mass Spectrometry (Compact PTR-TOF-MS 1000, Ionicon, Austria) to identify and quantify the spectrum of volatile organic compounds (VOCs).

SUMMARY:
This study aims to develop a non-invasive diagnostic method for metabolic syndrome (MetS) and metabolically healthy obesity (MHO) through analysis of exhaled air. Using proton-transfer-reaction mass spectrometry combined with machine learning algorithms, we will characterize volatile organic compound profiles in 300 participants across three groups: MetS patients, MHO patients, and healthy controls. The primary goal is to create and validate a classification model capable of accurately differentiating these metabolic states based on breath analysis.

DETAILED DESCRIPTION:
This study focuses on characterizing the volatilome - the complete set of volatile organic compounds in exhaled air - as a novel biomarker source for metabolic health assessment.

The study represents the first comprehensive attempt to compare volatilome signatures between metabolically healthy and unhealthy obesity phenotypes. Successful validation of this approach could establish breath analysis as a new diagnostic paradigm in metabolic medicine, enabling rapid, non-invasive screening and personalized treatment strategies for patients with obesity-related conditions.

Methodological innovations include real-time breath analysis capabilities and development of specialized machine learning algorithms for pattern recognition in complex mass spectrometry data. The findings are expected to contribute significantly to understanding metabolic pathway alterations in different obesity phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* For Group 1 (Metabolic syndrome): Age >18 years, signed informed consent, diagnosis of Metabolic Syndrome (IDF 2006 criteria: waist circumference >94 cm (men)/ >80 cm (women) + ≥2 of: BP ≥130/85 mmHg or antihypertensive therapy; TG ≥1.7 mmol/L; HDL-C <1.03 mmol/L (men) / <1.29 mmol/L (women); Fasting glucose ≥5.6 mmol/L).
* For Group 2 (Metabolically healthy obesity): Age >18 years, signed informed consent, waist circumference ≥94 cm (men) / ≥80 cm (women), absence of other Metabolic Syndrome criteria (hypertension, dyslipidemia, impaired fasting glucose).
* For Group 3 (Control): Age >18 years, signed informed consent, normal BMI, absence of signs of Metabolic Syndrome.

Non-inclusion criteria for all groups:

* Inability to provide informed consent;
* History of myocardial infarction or stroke;
* Chronic kidney disease stage 3B, 4, 5 (eGFR <30 ml/min/1.73m2);
* Acute or subacute cardiovascular disease;
* Familial hypercholesterolemia;
* Bronchopulmonary diseases;
* Acute or chronic infectious diseases;
* Type 1 or Type 2 diabetes mellitus;
* Systemic connective tissue diseases;
* Current or past history of oncological diseases;
* Severe liver dysfunction, decompensated liver cirrhosis (Child-Pugh class C);
* Pregnancy or lactation;
* Severe mental illness (severe dementia, schizophrenia);
* Comorbid conditions with life expectancy less than 1 year.

Exclusion Criteria:

* Patient refusal to continue participation in the study;
* Identification of any non-inclusion criteria after enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults (≥18 years) from three groups: 1) Patients with Metabolic Syndrome (IDF, 2005 criteria), 2) Patients with metabolically healthy obesity (BMI≥30, no metabolic abnormalities), and 3) Healthy controls (BMI<25, no metabolic disorders).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Specificity of the combined PTR-MS and machine learning model. | Through study completion, after all participant samples are collected and the final model is validated (anticipated within 1 year).
  Specificity (true negative rate) of the diagnostic model, based on the analysis of exhaled breath VOCs by PTR-MS and subsequent machine learning classification, for distinguishing between participants with Metabolic Syndrome, Metabolically Healthy Obesity, and healthy controls. The value will be reported with a 95% confidence interval.
Sensitivity of the combined PTR-MS and machine learning model. | Through study completion, after all participant samples are collected and the final model is validated (anticipated within 1 year).
  Sensitivity (true positive rate) of the diagnostic model, based on the analysis of exhaled breath Volatile Organic Compounds (VOCs) by Proton Transfer Reaction Mass Spectrometry (PTR-MS) and subsequent machine learning classification, for distinguishing between participants with Metabolic Syndrome, Metabolically Healthy Obesity, and healthy controls. The value will be reported with a 95% confidence interval.
Area Under the Receiver Operating Characteristic Curve (AUC-ROC) of the combined PTR-MS and machine learning model. | Through study completion, after all participant samples are collected and the final model is validated (anticipated within 1 year).
  The Area Under the Receiver Operating Characteristic Curve (AUC-ROC) as a composite measure of the diagnostic performance of the model based on PTR-MS breath analysis and machine learning. The AUC will be calculated for pairwise comparisons between the three study groups (Metabolic Syndrome vs. Metabolically Healthy Obesity; Metabolic Syndrome vs. Control; Metabolically Healthy Obesity vs. Control) and reported with a 95% confidence interval.

SECONDARY OUTCOMES:
Identification of specific Volatile Organic Compound (VOC) patterns. | Through study completion, after mass spectrometric data processing and database search are completed (anticipated within 1 year).
  Qualitative and quantitative assessment of specific Volatile Organic Compounds (VOCs) and VOC profiles significantly associated with Metabolic Syndrome and Metabolically Healthy Obesity compared to the control group. The identification of molecules will be performed using the Human Metabolome Database (HMDB) with an accuracy of ± 100 ppm.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital №1, Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
IPD will not be available for public sharing. The local Ethics Committee and national data protection laws do not permit public deposition of individual patient data. The informed consent does not include such provisions.